CLINICAL TRIAL: NCT03202121
Title: Relationship of Nocturnal Concentrations of Melatonin, γ-aminobutyric Acid and Total Antioxidants in Peripheral Blood With Insomnia After Stroke: Study Protocol for a Prospective Single-center Randomized Controlled Clinical Trial
Brief Title: Relationship of Nocturnal Concentrations of Melatonin, γ-aminobutyric Acid and Total Antioxidants With Insomnia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Rehabilitation Research Center (Other Government)
Responsible Party: Principal Investigator, Wei Zhang, Principal Investigator, China Rehabilitation Research Center
Other Study IDs: ChinaRRC_01
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- insomnia group: After screening according to inclusion and exclusion criteria, patients were assigned to insomnia group that contained 25 cases.
  Interventions: Other: insomnia group
- non-insomnia group: After screening according to inclusion and exclusion criteria, patients were assigned to non-insomnia group that contained 25 cases.
  Interventions: Other: non-insomnia group
- normal control: persons without stroke or insomnia served as normal controls that contained 25 cases.
  Interventions: Other: normal control

INTERVENTIONS:
Other: insomnia group — After screening according to inclusion and exclusion criteria, patients were assigned to insomnia group that contained 25 cases.
  Groups: insomnia group
Other: non-insomnia group — After screening according to inclusion and exclusion criteria, patients were assigned to non-insomnia group that contained 25 cases.
  Groups: non-insomnia group
Other: normal control — Persons without stroke or insomnia served as normal controls that contained 25 cases.
  Groups: normal control

SUMMARY:
To analyze the relationship of nocturnal concentrations of melatonin, γ-aminobutyric acid and total antioxidants with insomnia after stroke.

DETAILED DESCRIPTION:
Sleep disturbance, especially insomnia, is a common complication after ischemic stroke for the patients during rehabilitation of cerebral infarction. Actually, more than half of ischemic stroke patients have insomnia complaints. Meanwhile, poor quality of sleep may greatly impede stroke rehabilitation and induce other complications. Thus, it is of importance to study the insomnia for the post-stroke patients, especially when they are during rehabilitation of cerebral infarction.

Melatonin is a pineal hormone with the peak nocturnal secretion. Melatonin typically takes a large responsibility in coordination with the circadian rhythms and further serves as a regulator in the sleep function. The secretion peak of melatonin is around midnight to 3:00 a.m.. Along with other antioxidants, the melatonin can also work as an effective neuroprotective enzyme against neurodegeneration and ischemic brain injury. Thus, the melatonin is known to take an important role in acute ischemic stroke, with a rhythm impairment and nocturnal decrease. γ-Aminobutyricacid (GABA) is likewise a strong sleep regulator that may activate GABA receptors as well as inhibitors of waking processes. It is known that GABA level in the human body is strongly associated with the impairment of patients in the acute ischemic stroke. Antioxidant may take a critical role in the balance of oxidation by scavenging free radicals, so it is regarded as an important marker in studying the insomnia for the post-stroke patients. However, to our knowledge, there is almost no report on simultaneous measurements of levels of melatonin, GABA and antioxidants in the bloods of patients during the convalescence of ischemic stroke or on studying their association with the insomnia complication for the post-stroke patients.

Therefore, this prospective single-center randomized controlled clinical trial was designed to investigate the relationship of nocturnal concentrations of melatonin, γ-aminobutyric acid and total antioxidants with insomnia after stroke by comparing the nocturnal concentrations of melatonin, GABA and total antioxidants in stroke patients with insomnia or without insomnia and normal controls.

Data management Clinical researchers accurately, completely, timely filled out the clinical trial observation form. Data were recorded electronically by data managers using a double-data entry strategy. The electronic database was locked by the project manager after checking. All data were analyzed statistically by professional statisticians. Anonymized trial data will be published at www.figshare.com.

Statistical analysis Data were presented as the mean ± standard deviation for normally distributed variables, or median values (P25, P75) for non-normally distributed variables. Student's t-tests or nonparametric Mann-Whitney tests were performed to compare the differences between normally distributed variables or non-normally distributed variables. For the analysis of biochemical test results, data were transferred to normal distribution and Hotelling's T2 tests were performed. Before entering variables into the regression model, centering predictor variables were performed to avoid nonessential collinearity. Binary logistic regression analysis was conducted to identify the association between variables or variables interaction and insomnia diagnosis after infarction. Multiple linear regression analysis was carried out to determine the correlation between variables or variables interaction and sleep-related scores, such as Epworth Sleepiness Scale scores, Pittsburgh Sleep Quality Index scores, Insomnia Severity Index scores, Morningness-Eveningness Questionnaire (Chinese version) scores and Fatigue Severity Scale scores by using backward method. P values < 0.05 were considered statistically significant. SPSS 22.0 software was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Infarction occurred in the middle cerebral artery blood supply area (Identified by medical record, magnetic resonance imaging, magnetic resonance angiography, computed tomography or computed tomography angiogram)
* Diagnostic criteria for insomnia of Diagnostic and Statistical Manual of Mental Disorders (4th edition)
* Course of disease ≥ 3 months
* Mini-Mental State Examination > 27
* Age ranged from 50 to 70 years old
* Right handedness

Exclusion Criteria:

* Cognitive and language disorders
* History of rheumatism, cancer, severe liver and kidney dysfunction, benign prostatic hyperplasia, and severe cardiac insufficiency, besides hypertension, diabetes, and coronary atherosclerotic heart disease
* High-risk sleep apnea, i.e., STOP-Bang Questionnaire ≥ 3
* Unexplained limb pain, many times of getting up in the night to urinate or restless legs syndrome
* Frequency of application of sleeping drugs > once/week or the use of psychotropic drugs, such as anti-anxiety and depression drugs, and antipsychotic drugs
* Frequency of drinking coffee and other stimulating drinks > three times/week
* Drug or alcohol abuse
* Insomnia caused by poor sleeping conditions, such as noise, light, and bedmate interference
* Insomnia before affecting stroke
* Hamilton Depression Scale > 20 or Hamilton Anxiety Scale > 14
* Participation in other clinical trials

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This is a prospective single-center randomized controlled clinical trial in the China Rehabilitation Research Center. Stroke patients during rehabilitation have been recruited since July in 2014. After screening according to inclusion and exlcusion criteria, patients were assigned to insomnia group and non-insomnia group. Simultaneously, persons without stroke or insomnia served as normal controls. Each group contained 25 cases.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Nocturnal concentrations of melatonin | 1 day at 3:00 a.m
  Melatonin is a pineal hormone with the peak nocturnal secretion. Melatonin typically takes a large responsibility in coordination with the circadian rhythms and further serves as a regulator in the sleep function. The secretion peak of melatonin is around midnight to 3:00 a.m.. Along with other antioxidants, the melatonin can also work as an effective neuroprotective enzyme against neurodegeneration and ischemic brain injury. Thus, the melatonin is known to take an important role in acute ischemic stroke, with a rhythm impairment and nocturnal decrease.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale | 1 day at 3:00 a.m
  A tool used for quantifying stroke severity. The full score is 42. High score suggests severe nerve injury.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Ph.D, Principal Investigator — China Rehabilitation Research Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang W, Li F, Zhang T. Relationship of nocturnal concentrations of melatonin, gamma-aminobutyric acid and total antioxidants in peripheral blood with insomnia after stroke: study protocol for a prospective non-randomized controlled trial. Neural Regen Res. 2017 Aug;12(8):1299-1307. doi: 10.4103/1673-5374.213550. PMID 28966645